CLINICAL TRIAL: NCT01889875
Title: Immunological Comparison of AIT and SCIT Immunotherapy Against Grass Pollen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: ALK-Abelló A/S (Industry)
Responsible Party: Principal Investigator, Vibeke Backer, Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Graesallergi
Record Dates: First submitted 2013-06-24; First posted 2013-07-01 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Allergic Rhinitis Due to Grass Pollens

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (No Intervention)
- Subcutaneous Immunotherapy (SCIT) (Active Comparator): Treatment using ALK AluTard 225 "Phleum pratense"
  Interventions: Drug: ALK AluTard 225 "Phleum pratense"
- Sublingual Allergen Immunotherapy Tablets (AIT) (Active Comparator): Treatment using ALK Grazax 75,000 SQ-T "Phleum pratense"
  Interventions: Drug: ALK Grazax 75,000 SQ-T "Phleum pratense"

INTERVENTIONS:
Drug: ALK Grazax 75,000 SQ-T "Phleum pratense"
  Arms: Sublingual Allergen Immunotherapy Tablets (AIT)
Drug: ALK AluTard 225 "Phleum pratense"
  Arms: Subcutaneous Immunotherapy (SCIT)

SUMMARY:
Treatment of pollen allergies can be roughly divided into symptomatic treatment (e.g. antihistamines, steroids) and potentially curative immunotherapy. Immunotherapy can be delivered using subcutaneous or oral (mucosal) routes, with similar clinical outcome. The study seeks to compare immunological changes during subcutaneous (SCIT) and sublingual tablet (AIT) immunotherapy of grass pollen allergy (hayfever).

DETAILED DESCRIPTION:
Worldwide, more than 400 million people have allergic rhinitis, and sick-leave due to this condition costs societies billions of dollars annually1. Allergic rhinitis is most commonly treated with oral antihistamines and intranasal corticosteroids2. For moderate-severe rhinitis with poor control on topical treatment, immunotherapy should be considered3. Allergen immunotherapy is the only disease-modifying treatment available for IgE mediated allergy.

Immunotherapy is most commonly administered with subcutaneous injections of SQ-standardized allergen extracts (SCIT) and to a lesser extent, as sublingual drops (SLIT). However, other options now exist with the newly developed sublingual allergen immunotherapy tablets (AIT). The clinical effect of AIT4 and SCIT5 against grass pollen allergy has been demonstrated in large double-blind-placebo-controlled registration trials. These studies report significant reductions of symptom scores (AIT 30%, SCIT 32%) and seasonal rescue medication scores (AIT 38%, SCIT 41%) when compared with placebo4,5, persisting several years after withdrawal4,6. Immunotherapy may prevent new sensitizations and progression of rhinitis to asthma7-11. Allergen immunotherapy is generally well tolerated with few side effects, although a potential risk of anaphylactic reactions exists 12. A review of recent parallel meta-analyses on immunotherapy for grass pollen rhinitis suggests that the safety profile of AIT is superior to that of SCIT13.

The recommended length of immunotherapy with both SCIT and AIT is 3-5 years2, although the route of administration and the doses of allergen differ substantially. SCIT involves an up-dosing phase lasting 12-15 weeks with one or more weekly injections of increasing doses of allergen followed by a maintenance dose every 6-10 weeks. AIT starts with the daily maintenance dose, resulting in high cumulative doses. It is largely unknown whether the immunological mechanisms involved in the clinical effect are the same.

The changes in immunology have been extensively investigated for SCIT, and the most pronounced patterns are: 1) the induction of blocking antibodies, 2) a shift in Th1/Th2 balance towards Th1, and 3) induction of regulatory T cells. Similar mechanisms seem to be in play for AIT 14-16. Increases in allergen-specific non-IgE antibodies have been demonstrated in large trials of both SCIT and AIT treatment17,18, and studies have demonstrated that serum antibodies can reduce in vitro reactions mimicking allergic responses, such as IgE binding to allergen, IgE facilitated antigen presentation and basophil activation19-22, suggesting that both humoral and cellular effects play a role23.

The aim of the present study was to compare the effect of AIT and SCIT on antibody titers (IgE and IgG4), on allergen-IgE interaction in competition assays (IgE-blocking factor and FAP inhibition) and on effector cell activation (BAT). Nasal challenges were included to assess the changes in nasal response to grass pollen allergen.

ELIGIBILITY:
Inclusion Criteria:

* history of rhinitis with hay fever symptoms during the grass pollen season,
* a skin-prick-test-verified grass pollen allergy (Phleum pratense),
* eligibility for immunotherapy based on ARIA guidelines

Exclusion Criteria:

* current long-term systemic steroid treatment,
* previous immunotherapy,
* asthma and outside-season airway hyperresponsiveness (AHR) (September 2011),
* pregnancy,
* negative RAST for grass, and
* treatment side effect

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Changes over time in specific Antibodies | 0, 1, 2, 3, 6, 7, 10, 12, and 15 months post treatment start
  IgE, IgG4
Changes over time in Basophil Activation Test | 0, 1, 3, 6, 7, 10, 12, and 15 months post treatment start

SECONDARY OUTCOMES:
Changes over time in Nasal Challenge symptoms | 0, 3, 10, and 15 months post treatment start

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg University Hospital, Copenhagen NV, Denmark, Denmark

REFERENCES:
- [Derived] Aasbjerg K, Backer V, Lund G, Holm J, Nielsen NC, Holse M, Wagtmann VR, Wurtzen PA. Immunological comparison of allergen immunotherapy tablet treatment and subcutaneous immunotherapy against grass allergy. Clin Exp Allergy. 2014 Mar;44(3):417-28. doi: 10.1111/cea.12241. PMID 24734285